CLINICAL TRIAL: NCT04108806
Title: Study of Peripheral Arterial Calcification as a Possible Predictor of Outcome After Endovascular Therapy
Brief Title: Study of Peripheral Arterial Calcification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, hazem mohamed zaki mohamed, Resident of vascular surgery, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Endovascular therapy in PAC
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: PAD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovascular therapy (Experimental): Outcome of endovascular therapy on PAC
  Interventions: Procedure: Endovascular therapy

INTERVENTIONS:
Procedure: Endovascular therapy — Ballon dialtation of the diseased artery

SUMMARY:
Aim of the work :

1. Using different calcification scoring systems to investigate the association between arterial calcification and clinical outcome following endovascular therapy

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a worldwide health problem and its prevalence is increasing among aging population. Symptomatic PAD Is a major cause of major amputation with reduction of the functional capacity and quality of life . Arterial calcification is calcium crystallization deposits in the extracellular matrix of the intima and media . Medial calcification is usually associated with chronic kidney disease and diabetes mellitus, while intimal calcification comes usually as a part of atherosclerotic process . The relationship between calcification and PAD is well established . Arterial calcification is associated with increased risk of procedural failure and major amputation . Many calcium scoring systems have been proposed, including peripheral arterial calcium scoring scale (PACSS which highlights the pathologic location of calcification along with the length of the segment affected. The peripheral academic research consortium (PARC) suggested another calcium scoring scale that classified calcification into 4 major grades . The DEFENETIVE Ca++ have proposed another calcium severity scoring . Intravascular Ultrasound (IVUS) is highly sensitive to presence and location of atherosclerotic calcium .

The impact of intimal and medial vascular calcification on the safety and effectiveness of endovascular devices to treat symptomatic peripheral arterial disease (PAD) remains poorly defined warranting continued research to elaborate relationship between calcification and endovascular outcome.

ELIGIBILITY:
Inclusion Criteria:

1. patients with peripheral arterial disease
2. patients with disabling limb claudication
3. patients with rest pain
4. patients with minor tissue loss
5. patients admitted to vascular surgery department for endovascular intervention of a denovo lower limb arterial lesion

Exclusion Criteria:

* 1)Patient's age less than 50. 2)Patients with major tissue loss [ Rutherford category 6] 3)Patients with recurrent lesion after previous intervention. 4)Patients with double level arterial lesion. 5) Patients refusing to participate in this study

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-27 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09-27 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 1 year
  which means maintaining vessel patency without restenosis or need for re-intervention.
Major adverse limb events (MALE): | 1year
  by which we mean repeated endovascular therapy, surgical revision, or major amputation during follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Elsayed, Study Director — Assiut University; Ayman Sayed, Principal Investigator — Assiut University

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22107687/